CLINICAL TRIAL: NCT03961581
Title: Effectivness of Distraction by Electric ride-on Cars for Peri Operative Anxiety in Ambulatory Pediatric Surgery: a Randomised Controlled Study
Brief Title: Effectivness of Distraction by Electric ride-on Cars for Peri Operative Anxiety in Ambulatory Pediatric Surgery
Acronym: PTIBOLID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-02
Record Dates: First submitted 2019-04-11; First posted 2019-05-23 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- car (Experimental): Children who will use cars to go from the double-door entrance of the block to the operative room.
  Interventions: Behavioral: Using electric car
- bed (No Intervention): Children who will use bed to go from the double-door entrance of the block to the operative room.

INTERVENTIONS:
Behavioral: Using electric car — Child will use little electric cars to go to the reception of operating theatre to operating room.
  Arms: car

SUMMARY:
The main objective of this study is to measure perioperative anxiety in children from 2 to 10 years old in two distinct homogeneous groups before and after the ride in electric cars versus bed travel in the operating room.

The secondary objectives will be to measure the anxiety at the induction, the pain and the agitation of the children in SSPI as well as the satisfaction and the lived experience of the parents during the ambulatory stay of their child in the two groups journey in electric cars versus trip in bed.

It is a prospective, randomized, single-centric observational study (small electric cars versus bed-ridden), focusing on children during their stay in the operating theater at the CHU Nord of Marseille for ENT and ophthalmic surgery.

This study on the use of electric cars as a means of locomotion within the block may lead to other multicenter studies.

DETAILED DESCRIPTION:
Peri operative anxiety is one of major issues of pediatric anesthesia. Our efforts to decrease children anxiety improve pain, agitation ans behavioral changes during post operative period. Guidelines in pediatric anesthesia are to take into account anxiety in order to enhance recovery after anesthesia and to develop ambulatory surgery.

Pharmacological and non pharmacological tools are used. Midazolam is a benzodiazepin widely used but its indesirable effects such as paradoxical reactions, prolonged sedation and adverse behavioral changes are a brake to enhance recovery after anesthesia programs. Non pharmacological procedures are more promising (parental presence, behavioral preparation programs and distraction) but their etablishment is time consuming, requiring teaching programs, and changing habits. To our knowledge, distraction with ride-on car has not been studied yet.

Little electric car can carry children aged 2 years and more, it can be driven by children under adult distant command. Weight is limited to 35 kg (x pounds). Our hospital has 3 differents car models which allow children to choose for their prefered one et to become part of the adventure. Parental separation could be favored by this device.

Surgical procedures are ophtalmologic and oto rhino laryngologic, in an ambulatory ward receiving children ASA 1 to 3. Anesthesic procedure is the same for every child, inhalatory induction with sevoflurane following by perfusion for morphinic administration and oral intubation. To note, premedication is avoided and replaced by important information and reinsurrance of parents.

Chlidren will be randomised by block every week to go to operating room using gurney (goup a) or ride-on electric car (group b). Primary outcome is peri operative pediatric anxiety measured by Yale validated scale (m-YPAS). Other outcomes concern post opérative period (anxiety, pain, agitation), parental lived and satisfaction.

PTIBOLID is a monocentric prospective randomised controlled open study wich will include 110 patients in hopital Nord, Marseille, AP-HM.

ELIGIBILITY:
Inclusion Criteria:

* Children operated in ENT and ophtalmology
* Max 35 kg (advice from little electric car manufacturer)
* 2 years old minimum (psychomotor coordination)
* 10 years old maximum
* Ambulatory unit

Exclusion Criteria:

* < 2 years old
* Cognitive and physical impairment that forbids the use of cars
* Refusal of cooperation of the child
* Emergency surgery
* Consent of one of the parents for the study
* Refusal of cooperation of the parents
* Lack of understanding of the study

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Peri operative anxiety | 30 minutes
  Perioperative anxiety measured by the Modified Yale Preoperative Anxiety Scale (mYPAS )questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier ARNAUD, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Pastene B, Piclet J, Praud C, Garcia K, Louis K, Schmidt C, Boyadjiev I, Boucekine M, Baumstarck K, Bezulier K, Bouvet L, Zieleskiewicz L, Leone M. Pre-operative distraction using electric ride-on cars for children undergoing elective ambulatory surgery: A randomised controlled trial. Eur J Anaesthesiol. 2023 Mar 1;40(3):190-197. doi: 10.1097/EJA.0000000000001758. Epub 2022 Oct 3. PMID 36204923